CLINICAL TRIAL: NCT01857726
Title: A Randomized Open Label Pilot Study Comparing Transarterial Chemoembolization Versus Transarterial Chemoembolization/Transarterial Chemoinfusion Combination in Advanced Hepatocellular Carcinoma With Portal Vein Invasion
Brief Title: Comparison of TACE Versus TACE/TACI Combination in Advanced Hepatocellular Carcinoma With Portal Vein Invasion
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants were enrolled
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jung-Hwan Yoon, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PVT_TACE/TACI
Record Dates: First submitted 2013-05-13; First posted 2013-05-20 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; portal vein invasion; transarterial chemoembolization; transarterial chemoinfusion
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Doxorubicin; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- The TACE/TACI combination group (Experimental): Transarterial chemoembolization with doxorubicin/transarterial chemoinfusion with cisplatin combination
  Interventions: Drug: Doxorubicin; Drug: Cisplatin
- The TACE-only group (Active Comparator): Transarterial chemoembolization with doxorubicin
  Interventions: Drug: Doxorubicin

INTERVENTIONS:
Drug: Doxorubicin — Transarterial chemoembolization (TACE) with adriamycin
  Other Names: Adriamycin
Drug: Cisplatin — transarterial chemoinfusion with cisplatin 50-100 mg
  Arms: The TACE/TACI combination group

SUMMARY:
The aim of this study is to compare the efficacy of transarterial chemoembolization with adriamycin to transarterial chemoembolization with adriamycin/transarterial chemoinfusion with cisplatin combination in advanced hepatocellular carcinoma with portal vein invasion.

DETAILED DESCRIPTION:
Potentially curative treatments for hepatocellular carcinoma (HCC) include surgical resection, liver transplantation, and local ablative therapy.

However, HCC patients are diagnosed at advanced stages in Korea. Especially, HCCs with portal vein invasion are unresectable and they are not suitable for other curative therapies. For these patients, the optimal treatment remains largely controversial. As a palliative treatment, the benefit of transarterial chemoembolization (TACE) had been shown in patients with unresectable HCC and without portal vein invasion by several trials. In patients with main portal vein invasion, TACE is theoretically contraindicated because of the potential risk of hepatic failure resulting from ischemia after TACE. However, recent studies have revealed that TACE could safely be performed in these patients.

The aim of this study is to compare the efficacy of transarterial chemoembolization (TACE) with adriamycin to transarterial chemoembolization with adriamycin/transarterial chemoinfusion (TACI) with cisplatin combination in advanced hepatocellular carcinoma with portal vein invasion.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical or histological diagnosis of HCC based on the guidelines of the AJCC
* Patients with advanced HCC with invasion of major branch(es) of portal vein in the arterial phase of dynamic CT or MRI
* Patients who have received previous local therapy treatments (RFA, PEI, cryoablation, surgery, resection) are eligible
* Age : 18 years to 80 years
* ECOG Performance Status of 0 to 2
* Child-Pugh class A (Child-Pugh score 5-6)
* Adequate bone marrow, liver function as assessed by the following laboratory requirements to be conducted within 7 days prior to screening:

  * WBC count > 2,000/mm3
  * Absolute neutrophil count > 1,000/mm3
  * Hb ≧ 8.0 g/dL
  * Platelet count ≧ 50,000 /mm3
  * Bilirubin ≦ 3 mg/dL
  * Adequate clotting function: INR < 2.3 or < 6sec

Exclusion Criteria:

* Child-Pugh score ≧ 7
* ECOG Performance Status ≧ 3
* Patients with chronic kidney disease or serum creatinine ≥ 1.2 mg/dL
* History of organ allograft
* Patients with uncontrolled co-morbidity which needs treatment
* Patients who have received prior systemic chemotherapy
* Patients with extrahepatic metastasis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-07; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival | every 12 weeks, up to 48 weeks

SECONDARY OUTCOMES:
Time-to-progression | every 12 weeks, up to 48 weeks
Progression-free survival | every 12 weeks, up to 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Hwan Yoon, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea